CLINICAL TRIAL: NCT04056897
Title: International Multicenter, Randomized, Double-blind, Double-masked, Placebo-controlled Study of the Efficacy and Safety of BCD-132 Using an Active Reference Drug (Teriflunomide) for the Treatment of Patients With Multiple Sclerosis
Brief Title: Comparative Study of the Efficacy and Safety of BCD-132 With Teriflunomide and Placebo in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-132-2
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-132, 125 mg (Experimental): 72 patients
  Interventions: Biological: BCD-132, 125 mg
- BCD-132, 500 mg (Experimental): 72 patients
  Interventions: Biological: BCD-132, 500 mg
- Teriflunomide (Active Comparator): 72 patients
  Interventions: Drug: Teriflunomide
- Placebo (Placebo Comparator): 54 patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: BCD-132, 125 mg — IV infusion every 24 weeks in combination with placebo tablet daily. The total duration of blinded therapy is 100 weeks (a total of 5 cycles of therapy BCD-132 in combination with a daily placebo)
  Arms: BCD-132, 125 mg
Drug: Teriflunomide — 14 mg teriflunomide tablet. Per os. Daily in combination with IV placebo. The total duration of blinded therapy is 100 weeks (a total of 5 cycles of placebo IV therapy in combination with daily administration of teriflunomide)
  Arms: Teriflunomide
Drug: Placebo — intravenous infusion in combination with placebo tablet daily. The total duration of blinded therapy is 100 weeks
  Arms: Placebo
Biological: BCD-132, 500 mg — IV infusion every 24 weeks in combination with placebo tablet daily. The total duration of blinded therapy is 100 weeks (a total of 5 cycles of therapy BCD-132 in combination with a daily placebo)
  Arms: BCD-132, 500 mg

SUMMARY:
International multicenter, randomized, double-blind, double-masked, placebo-controlled study of efficacy and safety of BCD-132 (JSC BIOСAD, Russia) using an active reference drug (teriflunomide) for the treatment of patients with multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study;
2. Men and women aged from 18 to 60 years (inclusive) on the day of signing informed consent;
3. Confirmed diagnosis of relapsing-remitting multiple sclerosis (according to McDonald criteria 2017 revision);
4. Documentary evidence that within the last 12 months before signing informed consent the patient had:

   1. At least 1 relapse, or
   2. 2 relapses over the past 2 years, or
   3. At least 1 Gadolinium enhancing T1-weighted lesion and 1 relapse over the past 2 years (24 months) before signing informed consent;
5. The patient should be neurologically stable during 30 days before signing informed consent (i.e. the patient should not have any new or aggravated neurological symptoms, as told by the patient); or the patient's condition should be completely stabilized since the last relapse, and the duration of stabilization should be at least 30 days);
6. Total EDSS score of 0 to 5.5 inclusive;
7. The presence of immunoglobulins G antibodies to the Varicella-Zoster virus according to the results of screening examination;
8. The absence of suicidal ideation and suicidal behavior established in the screening, according to the C-SSRS score;
9. The willingness of patients of both sexes and their partners with preserved reproductive function must implement reliable contraceptive methods starting from signing informed consent, throughout the study and within 48 weeks after the last dose of the drug in this study. This requirement does not apply to patients after operative sterilization. Reliable contraception methods include one barrier method in combination with one of the following: spermicides, intrauterine device/oral contraceptives;

Exclusion Criteria:

1. Primary or secondary progressive MS;
2. The duration of the MS for more than 10 years with EDSS ≤ 2.0;
3. Other conditions (except for multiple sclerosis) that can affect the assessment of MS symptoms: to mask, aggravate, change symptoms of multiple sclerosis, result in clinical signs or laboratory instrumental findings suggesting multiple sclerosis;
4. A relapse during the screening period;
5. Systemic corticosteroids used within 30 days before signing informed consent;
6. Diseases requiring prolonged systemic therapy with corticosteroids and / or immunosuppressive drugs, with the exception of MS;
7. Any acute infections, relapses of chronic infections or any other chronic diseases that are present on the day of signing informed consent and can, as judged by the Investigator, negatively affect the patient's safety during the study treatment;
8. Congestive heart failure (Grade IV NYHA);
9. A history of ischemic cerebrovascular disease or spinal cord ischemia, myelopathy, neuromyelitis optica, sarcoidosis;
10. HIV, hepatitis B, hepatitis C, or syphilis;
11. Metabolic abnormalities (disorders) manifesting as:

    1. baseline creatinine levels increased more than 2-fold vs. upper limit of normal;
    2. baseline urea levels increased more than 3-fold vs. upper limit of normal;
    3. baseline ALT (Alanine aminotransferase), AST (Aspartate Aminotransferase) or GGT (Gamma-glutamyltransferase) levels increased more than 2.5-fold vs. upper limit of normal;
    4. baseline bilirubin levels increased more than 1.5-fold vs. upper limit of normal;
12. Baseline leukocyte counts lower than <3.0 × 109/L, platelet counts lower than <125 × 109/L or hemoglobin levels <100 g/L;
13. TSH (thyroid stimulating hormone) level increased more than 2-fold vs. upper limit of normal;
14. A history of severe depression, suicidal thoughts or suicide attempts ;
15. Pregnancy, lactation or planned pregnancy over the entire study period;
16. A history of use:

    * any time before signing informed consent: anti-B cell therapy drugs (rituximab, oсrelizumab, abatacept, belimumab, ofatumumab and others);
    * any time before signing informed consent: alemtuzumab, daclizumab, teriflunomide, mitoxantrone, cladribine, as well as total lymphatic irradiation (TLI), bone marrow transplantation;
    * within 2 years (24 months) before signing informed consent: cyclophosphamide, cyclosporine, azathioprine; mycophenolate mofetil, fingolimod and sphingosine-1-phosphate (S1P) receptor modulator, natalizumab;
    * immunoglobulin therapy within 30 days before signing informed consent.
17. Intolerance, including hypersensitivity to any of the components of BCD-132 / teriflunomide, premedication, as well as conditions that, as judged by the Investigator, are a contraindication to the appointment of the above drugs;
18. The history of severe allergic or anaphylactic reactions;
19. Progressive multifocal leukoencephalopathy (PML);
20. Known alcoholic or drug dependency or signs of present alcoholic/drug dependence that, in the Investigator's opinion, can be contraindications for study therapy of MS with anti-CD20 Mab or limit treatment compliance;
21. Inability to follow the Protocol procedures (in the Investigator's opinion);
22. Contraindications to MRI or use of gadolinium-containing contrast agents:

    1. Metal foreign objects in the body: magnetic implants, ferromagnetic clips for cerebral vessels, artificial heart valves, electronic middle ear implants, pacemakers;
    2. A history of allergy to gadolinium or gadolinium-containing contrast agents;
    3. Fear of cramped spaces; d) Kidney function impairment with a risk of delayed gadolinium elimination (creatinine level increased to more than 2 x upper limit of normal); d) Documented diagnosis of sickle cell or hemolytic anemia, hemoglobinopathy;
23. Any malignancies or a history of malignancies, except for cured basal cell carcinoma or cervical cancer in situ;
24. Vaccination within 4 weeks before signing informed consent (as told by the patient);
25. Participation in other clinical studies within 90 months before signing informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Number of T1 Gd+ Lesions (per scan) | week 24
  The number of T1 gadolinium enhancing (T1 Gd+) lesions

SECONDARY OUTCOMES:
CUA | week 24, week 100
  The number of combined unique active (CUA) lesions. Changes in MRI (magnetic resonance imaging) markers
Proportion of Patients Without Contrast-enhancing Lesions | week 24, week 100
  Changes in MRI markers
Number of New or Enlarging T2-weighted Lesions | week 24, week 100
  Changes in MRI markers
Number of Patients Without New or Enlarging T2-weighted Lesions | week 24, week 100
  Changes in MRI markers
Changes in T2-weighted Lesion Volume | week 24, week 100
  Changes in MRI markers
Changes in Hypointense T1-weighted Lesion Volume | week 24, week 100
  Changes in MRI markers
Whole-brain Volume Change according MRI | week 24, week 100
  Changes in MRI markers
Annual Average Frequency of Relapses | week 24, week 100
  Number of relapses during the year
Time to First Relapse | week 24, week 100
  Relapse-related variables
Number of Relapse-free Patients | week 24, week 100
  Relapse-related variables
Number of Patients With Sustained Disability Progression | week 24, week 100
  Relapse-related variables
Expanded Disability Status Scale (EDSS) | week 24, week 100
  EDSS is a scale for assessing neurologic impairment in MS. It consists of eight functional systems (FS) which are used to derive the EDSS steps (score) ranging from 0 (normal) to 10 (death due to MS). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Based on the assessment of each FS, the participant's score is determined between 0 to 10. A positive change from baseline indicates improvement
Timed 25-Foot Walk | week 24, week 100
  Quantitative mobility and leg function performance test based on a timed 25-walk.
9-Hole Peg Test (9 HPT) | week 24, week 100
  9HPT is a brief, standardized, quantitative test of upper extremity function
Symbol Digit Modalities Test (SDMT) | week 24, week 100
  SDMT it is neuropsychological test detecting not only the presence of brain damage, but also changes in cognitive functioning over time and in response to treatment.
36-Item Short Form Survey (SF-36) | week 24, week 100
  SF-36 it is a 36-item, patient-reported survey of patient health.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability
EQ-5D Questionnaire | week 24, week 100
  EQ-5D - European Quality of Life Questionnaire. It has two components: health state description and evaluation. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3.
MSQOL-54 Questionnaire | week 24, week 100
  MSQOL - Multiple Sclerosis Quality of Life-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores.
  MSQoL-54 has 0-100 scales. Higher values indicate better quality of life.
Number of Patients Who Developed AEs That, in the Investigator's Opinion, Are Related to Treatment | week 24, week 100
  The Proportion of Patients Who Developed AEs That, in the Investigator's Opinion, Are Related to Treatment
The Number of Patients Who Developed SAEs That, in the Investigator's Opinion, Are Related to Treatment | week 24, week 100
  SAE- Serious adverse event
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | week 24, week 100
  The Proportion of Patients, in Each Group, Who Developed СТСАЕ v. 5.0 Grade 3-4 AEs That, in the Investigator's Opinion, Are Related to Treatment CTCAE - Common Terminology Criteria for Adverse Events
The Number of Patients, in Each Group, Who Discontinued the Study Due to AEs/SAEs | week 24, week 100
  AE- adverse event, SAE - serious adverse event
Number of patients with binding and neutralizing antibodies | week 24, week 100
  The Proportion of binding and neutralizing positive patients
Beck Depression Inventory | week 24, week 100
  Beck Depression Inventory is a 21-item self-reporting questionnaire for evaluating the severity of depression. Minimum score -0, maximum score - 63.
  Higher total scores indicate more severe depressive symptoms.
C-SSRS | week 24, week 100
  The Columbia Suicide Severity Rating Scale, or C-SSRS, is a suicidal ideation and behavior rating scale.
  C-SSRS - Columbia-Suicide Severity Rating Scale. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. Assign a score of 0 if no ideation is present.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JSC BIOCAD
Locations (1):
- State Budgetary Healthcare Institution of Nizhny Novgorod region "Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod", Nizhny Novgorod, Russia